CLINICAL TRIAL: NCT02193113
Title: An Open Label, Single Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacodynamics of a Novel Intravitreal Plasma Kallikrein Inhibitor in Subjects With Central Involved Diabetic Macular Edema and Reduced Vision
Brief Title: A Phase I Single Ascending Dose Study of the Intravitreal Plasma Kallikrein Inhibitor KVD001 in Subjects With DME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KVD001-001
Record Dates: First submitted 2014-07-09; First posted 2014-07-17 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; DME; Plasma Kallikrein inhibitor; KVD001; KVD001-001; Intravitreal; IVT; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- KVD001 Injection Dose 1 (Experimental): Single 100 microliters (uL) intravitreal injection of KVD001 Injection Dose 1
  Interventions: Drug: KVD001 Injection
- KVD001 Injection Dose 2 (Experimental): Single 100uL intravitreal injection KVD001 injection Dose 2
  Interventions: Drug: KVD001 Injection
- KVD001 Injection Dose 3 (Experimental): Single 100uL intravitreal injection of KVD001 injection Dose 3
  Interventions: Drug: KVD001 Injection

INTERVENTIONS:
Drug: KVD001 Injection — A novel plasma kallikrein inhibitor
  Other Names: KVD001

SUMMARY:
This is a Phase 1 study to investigate the safety, tolerability of the novel plasma kallikrein inhibitor, KVD001 in subjects with diabetic macular edema. The study is the first step to investigate the hypothesis that plasma kallikrein plays an important role in the disease process behind diabetic macular edema in many patients

DETAILED DESCRIPTION:
The plasma kallikrein-kinin system has long been recognized as a key player in inflammatory processes, capillary leakage and angiogenesis in various organs. Recent work suggests that plasma kallikrein is central to the pathogenesis of Diabetic Macular Edema (DME) and that activation of the enzyme contributes to the excessive retinal vascular permeability leading to DME. Among different persons with DME, plasma kallikrein contributes both independently in some, and in association with Vascular Endothelial Growth Factor (VEGF) in others. However, the effect of plasma kallikrein appears to be independent of VEGF. Thus, growing scientific evidence points to plasma kallikrein inhibitors as an exciting potential new therapeutic opportunity directed at a novel VEGF-independent pathway that may reduce retinal vascular permeability and treat DME, in patients whose disease process is, at least in part, driven by the plasma kallikrein pathway.

This is an open label, single ascending dose study to investigate the safety, tolerability and pharmacodynamics of a novel plasma kallikrein inhibitor administered by intravitreal (IVT) injection in subjects with central involved diabetic macular edema and reduced vision.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult subjects 18 years of age and older
2. Confirmed diagnosis of Type I or Type II diabetes mellitus
3. Best corrected visual acuity, using Early Treatment Diabetic Retinopathy Study (ETDRS) electronic visual acuity (EVA) testing, of between 20/40 and 20/400 (Snellen equivalent) in the study eye
4. Fellow eye acuity 20/80 or better measured as above with no expectation of requirement for anti-VEGF treatment in fellow eye within 2 months of study drug administration
5. Presence of central involved DME in the study eye defined as Optical Coherence Tomography (OCT) Central Subfold Thickness (CST) ≥305 µm in women and ≥320 µm in men in the study eye
6. Subjects who fulfil one of the following criteria:

   1. Subjects who have not previously received an anti-VEGF treatment and who, in the view of the Investigator, can have initiation of anti-VEGF treatment in the study eye deferred for at least 2 months following the date of anticipated study drug administration
   2. Subjects who are receiving regular anti-VEGF intravitreal injections who:

      * Have received at least 3 intravitreal injections of an anti-VEGF treatment within the last 5 months (study drug administration will be at least 6 weeks after the most recent intravitreal administration of anti-VEGF) and
      * In the view of the Investigator, can have continuation of anti-VEGF treatment in the study eye deferred for at least 2 months following the date of anticipated study drug administration
   3. Subjects who have received anti-VEGF in the past (>3 months prior to study inclusion) but are not actively receiving treatment and who in the view of the Investigator, can have resumption of anti-VEGF or alternative treatment in the study eye deferred for at least 2 months following anticipated study drug administration
7. Subjects, who in the view of the Investigator, are not expected to require panretinal laser photocoagulation or intravitreal steroids or intraocular surgery in the study eye for at least 2 months following anticipated study drug administration
8. No prior treatment with panretinal photocoagulation or intravitreal steroid in the study eye within the previous 3 months
9. No prior treatment with systemic corticosteroids or systemic anti-VEGF therapy within the previous 3 months
10. Study participant voluntarily agrees to participate in this study and signs the Institutional Review Board (IRB) approved informed consent prior to performing any procedure

Exclusion Criteria:

1. Females who are pregnant or lactating, or expecting to become pregnant during the course of the study
2. Poorly controlled diabetes mellitus
3. Uncontrolled hypertension
4. Significant co-existing disease
5. Participation in an investigational intervention clinical study within 2 months prior to study inclusion
6. History of alcohol and/or drug abuse in the last 2 years
7. Men not willing to use appropriate birth control methods
8. Media clarity or pupillary dilation inadequate to obtain reasonable quality OCT and/or fundus image
9. Subjects employed by the Sponsor or in any relationship of dependence with the Sponsor and/or Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-07-18 (Actual); Primary Completion 2015-06-04 (Actual); Study Completion 2015-06-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a measure of safety and tolerability | 56 days

SECONDARY OUTCOMES:
Measurement of KVD001 plasma levels over time following intravitreal injection (with calculation of Tmax, Cmax, AUC and t1/2) | 28 days
Best Corrected Visual Acuity as measured by ETDRS EVA | 56 days

OTHER OUTCOMES:
Change in retinal thickness from baseline | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sun, MD, MPH, Principal Investigator — Joslin Diabetes Center; David Boyer, MD, Principal Investigator — Retina-Vitreous Associates Medical Group; Victor Gonzalez, MD, Principal Investigator — Valley Retina Institute, PA; Raj Maturi, MD, Principal Investigator — Midwest Eye Institute; Jack Wells, MD, Principal Investigator — Palmetto Retina Center
Locations (5):
- United States (5):
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Raj K. Maturi, MD PC, Indianapolis, Indiana
  - Beetham Eye Institute, Boston, Massachusetts
  - Palmetto Retina Center, West Columbia, South Carolina
  - Valley Retina Institute, PA, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's Website (KalVista Pharmaceuticals) — http://www.kalvista.com